CLINICAL TRIAL: NCT06033313
Title: Examining the Effect of Message Framing on Medication Beliefs, Intentions to Take Medications, Adherence to Medication, and Asthma Control Among College Students
Brief Title: Effects of Framing on Medication Beliefs, Intentions to Take Medication, Adherence, and Asthma Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Ruth Jeminiwa, Principal Investigator, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-221
Record Dates: First submitted 2023-06-14; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Asthma
Keywords: mHealth; message framing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positively framed text messages (Experimental): Positively framed text messages
  Interventions: Behavioral: Positively Framed text messages
- Negatively frame text messages (Experimental): Negatively framed text messages
  Interventions: Behavioral: Negatively Framed text messages

INTERVENTIONS:
Behavioral: Negatively Framed text messages — Negatively Framed text messages delivered to participants three times per week for 8 weeks.
  Arms: Negatively frame text messages
Behavioral: Positively Framed text messages — Positively Framed text messages delivered to participants three times per week for 8 weeks.
  Arms: Positively framed text messages

SUMMARY:
The goal of this study is to examine the effects of framed mobile messages on young adults' beliefs about their daily Inhaled Corticosteroids (ICS), intentions to take their ICS, adherence, and asthma control. College students (18-29 years) who owned a mobile phone and had a diagnosis of asthma with a prescription for an ICS will be recruited. Participants will be randomized to receive either gain- or loss-framed mobile messages three times per week for eight weeks. Outcomes including beliefs, intentions, adherence, and asthma control will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of asthma
* A prescription for an inhaled corticosteroid
* Enrolled in college
* Between 18-29 years of age
* Owns a mobile phone

Exclusion Criteria:

* Cannot read in english

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Asthma control | Data collection at baseline, week 4, and week 8
  Asthma control as measured by the Asthma Control Test (minimum value=5, maximum value= 25) Questionnaire (scores of 20 and above indicate asthma control)

SECONDARY OUTCOMES:
Changes in Medication Beliefs | Data collection at baseline and week 8
  Medication Beliefs as measured by the Beliefs about Medicines Questionnaire-Specific (This scale has two sub-scales : necessity (20- points) and concerns (20 points). A difference of necessity and concern scores shows the level of perceived necessity for the medication. Higher scores indicate higher perceived necessity for the medication.
Intentions to take medication as prescribed | Data collection at baseline and week 8
  Intentions to take inhaled corticosteroids as prescribed as measured by an intentions scale (minimum score = 3, maximum score = 15; higher scores indicate greater intentions; the scale was tested in the study)
Changes in Medication adherence | Data collection at baseline, week 4, and week 8
  Adherence to a daily dose of inhaled corticosteroid as measured by the Medication Adherence Report Scale for Asthma (MARS-A) (Minimum score = 10, maximum score = 50, higher scores indicate greater adherence)

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request
Supporting Information: Study Protocol, ICF
Time Frame: Immediately available upon request for the next 10-20 years
Access Criteria: This is not applicable